CLINICAL TRIAL: NCT02297334
Title: Reduction of Inflammation Reaction to Extracorporeal Circulation in Cardiac Surgery by Interleukin Dialysis
Brief Title: Removal of Cytokines During Extracorporeal Circulation in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANA-UKE-PV 4420
Record Dates: First submitted 2014-10-08; First posted 2014-11-21 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Coronary Artery Disease; Heart Valve Diseases
Keywords: CytoSorb(TM); cytokines; inflammation; cardiac surgery; extracorporeal bypass
MeSH Terms: conditions — Coronary Artery Disease; Heart Valve Diseases; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- With CytoSorb device (Active Comparator): Patients randomised to this arm are treated with the CytoSorb device during bypass.
  Interventions: Device: CytoSorb device
- Withouot device (No Intervention): Patients randomised to this arm are treated without the CytoSorb device during bypass.

INTERVENTIONS:
Device: CytoSorb device — In 20 patients the CytoSorb device will be installed into the extra corporeal circuit. A blood flow of 400ml/min is provided by an roller pump of the heart lung machine in a parallel stream to the main circulation.
  Other Names: polymer beads adsorbent
  Arms: With CytoSorb device

SUMMARY:
The aim of this study is to prove that using a CytoSorb(TM) filter in the cardiopulmonary circuit attenuates the inflammatory response to extracorporeal circulation in patients undergoing cardiac surgery. The hypothesis is that removing cytokines from patients' blood by the CytoSorb device significantly improves circulation and outcome in patients undergoing on-pump cardiac surgery.

DETAILED DESCRIPTION:
Cardiac surgery with cardiopulmonary bypass (CPB) induces an inflammatory response due to contact of patients' blood with foreign surfaces like tubes or the oxygenator, ischemic-reperfusion injury and surgical trauma. Inflammation is modulated by cytokines, especially, interleukins. The extent of cytokine release is further related to the duration of bypass and the amount of operating field suction. This results in a systemic inflammatory response syndrome (SIRS) with the risk of multiple organ dysfunction (MOD). Also in patients treated with extracorporeal membrane oxygenation (ECMO) an activation of the inflammation system is seen and accompanied with an increase of cytokine levels. The cytokine concentration correlates with the severity of the immune reaction and can be a predictor of the outcome of the patient. As severe SIRS and MOD significantly increase mortality, the attenuation of the inflammatory response is supposed to reduce morbidity and mortality after cardiac surgery.

For adult cardiac surgery and patients who are treated with an extracorporal assist device, a tool for cytokine elimination and attenuation of the inflammatory response seems to be beneficial.

In our study we are going to investigate if the use of the CytoSorb device can improve the outcome of patients undergoing elective coronar artery bypass and heart valve surgery.

ELIGIBILITY:
Inclusion Criteria:

* undergoing elective coronar bypass AND heart valve surgery
* expected duration of bypass more than 120 min

Exclusion Criteria:

* age under 18 years of age
* pregnancy
* medication that interacts with the immune system (e.g. steroids, immune suppressors)
* patients with diagnosed immunodeficiency (e.g. HIV/AIDS)
* heparin induced thrombocytopenia type II
* patients that decline participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-09; Primary Completion 2015-10 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Change of levels of cytokines during procedure compared to baseline | 1) 5 minutes before bypass 2) 2 hours after begin of bypass, 3) at the end of bypass, approximately 3 hours after begin of bypass, 4) 6 hours after bypass 5) 24 hours after bypass
  parameters to be measured are: interleukin (IL) 1, interleukin 6, interleukin 8, interleukin 10, tumor necrosis factor-alpha

SECONDARY OUTCOMES:
Change of hemodynamic parameters during procedure compared to baseline | 1) 5 kinutes before bypass 2) 2 hours after begin of bypass, 3) at the end of bypass, approximately 3 hours after begin of bypass, 4) 6 hours after bypass 5) 24 hours after bypass
  Hemodynamic and respiratory parameters such as mean arterial pressure, heart rate and peripheral oxygen saturation are recorded. In addition thermodilution parameters (stroke volume variability, global end diastole volume, extravascular lung water index, cardiac index, systemic vascular resistance) are measured. Volume and catecholamine therapies are managed by an algorithm based on thermodilution parameters.
Thromboelastometry | at the end of bypass, approximately 3 hours after begin of surgery
  At the end of extracorporeal circulation a rotation thromboelastometry analysis is performed and the clotting time (CT), the clot formation time (CFT), the maximum clot firmness (MCF) in In- and Ex-Tem and the MCF in Fib-Tem are measured. Based on an institutional algorithm the coagulation therapy is performed according to the results of the thromboelastometry.
Change of cognitive and emotional state in comparison to condition before surgery | 1)one day before surgery 2) 24 hours after bypass
  To evaluate, if the use of the cytokine-filter has any influence on cognitive function or the emotional state, the patients perform the mini-mental state examination and answer questions of the Geriatric Depression Scale questionaire. Results before and 24 hours after end of bypass are recorded.

OTHER OUTCOMES:
Amount of administered fluids | at the end of surgery, approximately 3 hours after begin of surgery
  The amount of fluids administered during operation is recorded.
Amount of administered catecholamines. | at the end of surgery, approximately 3 hours after begin of surgery
  The amount of catecholamines administered during operation is recorded.
Amount of administered catecholamines | after discharge from ICU, approximately 24 hours after surgery
  The amount of catecholamines administered during operation is recorded.
Change of a set of general laboratory parameters during procedure | 1) 5 minutes before bypass 2) 2 hours after begin of bypass, 3) at the end of bypass, approximately 3 hours after begin of surgery 4) 6 hours after bypass 5) 24 hours after bypass
  In laboratory tests we measure the whole blood count (red blood cells, white blood cells, thrombocytes), C-reactive protein, liver enzymes (GOT, GPT), kidney parameters (creatinine, glomerular filtration rate) and electrolytes (sodium, potassium, calcium) are measured.
Intensive care durations | after discharge from ICU, approximately 24 hours after admission
  After discharge from ICU the duration of stay and postoperative ventilation is recorded.
complication and adverse events | 24 hours after admission to ICU
  Any complications or adverse events, like death, bleeding, rethoracotomy or malignant arrhythmias are recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Jens C. Kubitz, MD PhD, Study Director — Department of Anaesthesiology Center of Anaesthesiology and Intensive Care Medicine University Medical Center Hamburg-Eppendorf University of Hamburg; Daniel A. Reuter, MD PhD, Study Chair — Department of Anaesthesiology Center of Anaesthesiology and Intensive Care Medicine University Medical Center Hamburg-Eppendorf University of Hamburg; Alexander März, MD, Principal Investigator — Department of Anaesthesiology Center of Anaesthesiology and Intensive Care Medicine University Medical Center Hamburg-Eppendorf University of Hamburg; Ingo Garau, MD, Principal Investigator — Department of Anaesthesiology Center of Anaesthesiology and Intensive Care Medicine University Medical Center Hamburg-Eppendorf University of Hamburg
Locations (1):
- Department of Anaesthesiology Center of Anaesthesiology and Intensive Care Medicine University Medical Center Hamburg-Eppendorf University of Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided